CLINICAL TRIAL: NCT03744702
Title: Pilot Study for Determining the Impact of Ascorbic Acid Treatment on the Development and Treatment of Vasodilation in Cardiac Surgery
Brief Title: Impact of Ascorbic Acid Treatment on the Development and Treatment of Vasodilation in Cardiac Surgery
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Erica D. Wittwer, M.D., Ph.D., Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-003358
Record Dates: First submitted 2018-11-14; First posted 2018-11-16 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Vasoplegia
Keywords: vasoplegia; cardiac surgery; ascorbic acid
MeSH Terms: conditions — Vasoplegia | interventions — Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): All patients will receive ascorbic acid as this is a pilot study.
  Interventions: Drug: Ascorbic Acid

INTERVENTIONS:
Drug: Ascorbic Acid — Patients will receive IV ascorbic acid.
  Other Names: Ascor

SUMMARY:
This is a prospective pilot study in which the effects of ascorbic acid administration are investigated in adult patients undergoing cardiac surgical procedures requiring cardiopulmonary bypass (CPB). Ascorbic acid (Vitamin C) is an essential cofactor in the biosynthesis of catecholamines, and critically ill patients are known to be ascorbate-deficient. In addition, cardiopulmonary bypass (CPB) decreases ascorbic acid concentrations. Cardiac vasoplegia is the loss of vascular tone despite adequate volume status and cardiac output, occurring commonly in patients after CPB. This necessitates the administration of vasopressors and alternative agents which can have deleterious effects. The administration of ascorbic acid to cardiac surgical patients may improve microcirculatory function, enhance endogenous catecholamine levels and decrease the need for exogenous vasopressor support.

DETAILED DESCRIPTION:
1. Specific Aims

The investigators aim to determine the feasibility of performing a study that can assess the impact of ascorbic acid administration on the development and severity of cardiac vasoplegia in cardiac surgical patients undergoing procedures at high risk for vasoplegia.

Specific Aim 1: Determine the feasibility of administration of high dose intravenous ascorbic acid in the operative and post-operative environments as well as sample size for a prospective, randomized, placebo controlled study.

Specific Aim 2: Determine baseline ascorbic acid plasma levels in a small cohort of cardiac surgical patients.

Specific Aim 3: Determine the impact of ascorbic acid administration on microvasculature as measured by dark field microscopy.

ELIGIBILITY:
Inclusion criteria:

* 18 years of age or older
* Undergoing cardiac surgery with the use of cardiopulmonary bypass
* Undergoing myectomy or valve replacement/repair

Exclusion criteria:

* Coronary artery bypass grafting (CABG)
* Circulatory arrest
* Active infection or sepsis
* Severe hepatic disease or ascites
* Pre-operative renal dysfunction requiring dialysis
* Pre-operative midodrine
* Pre-operative oral or intravenous steroid use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-06-28 (Actual); Primary Completion 2021-02-05 (Actual); Study Completion 2021-02-05 (Actual)

PRIMARY OUTCOMES:
Vasopressor duration in hours | Up to 10 days following surgery
  Total duration of vasopressor therapy
Vasopressor dose | Up to 10 days following surgery
  Total dose of vasopressor in norepinephrine equivalents (mcg)

CONTACTS AND LOCATIONS:
Overall Officials: Erica D Wittwer, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wieruszewski PM, Radosevich MA, Nei SD, Kashani KB, Normand SE, Schaff HV, Wittwer ED. Ascorbic acid and microcirculation in cardiothoracic surgery: a pilot feasibility trial and matched cohort study. J Cardiothorac Surg. 2025 May 22;20(1):234. doi: 10.1186/s13019-025-03486-8. PMID 40400032
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials